CLINICAL TRIAL: NCT03085953
Title: Study for the Employment Retention of Veterans
Acronym: SERVe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Portland State University (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Leslie Hammer, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: W81XWH-13-2-0020
Record Dates: First submitted 2017-02-15; First posted 2017-03-21 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Well-Being; Health Behavior; Workplace Outcomes
Keywords: Psychological health; Well-being; Employee
MeSH Terms: conditions — Health Behavior; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: Supervisor Intervention (Experimental): Supervisors in the intervention group will go through the Veteran Supervisor Supportiveness Training.
  Interventions: Behavioral: Veteran Supportive Supervisor Training
- Waitlist Control Group (Other): Supervisors will receive intervention following all measurement points, to serve as a waitlist control comparison group
  Interventions: Other: Waitlist Control

INTERVENTIONS:
Behavioral: Veteran Supportive Supervisor Training — The family supportive supervisor behavior (FSSB) training intervention developed by Hammer and colleagues (2011) will be used as the basis for the development of the VSST intervention in the present study. In addition, we will draw on critical elements of training provided by the Employer Support of the Guard and Reserve (ESGR), information about potential mental and physical health effects of being in combat, and information to help reduce the stigma associated with returning veterans; in other words, "de-clinicalizing" their symptoms. Furthermore, this intervention study falls under the more general rubric of soldier resilience, but more specifically addresses both veteran and family resilience upon return from combat. The details of the training content will be researched and developed during the funded project period.
  Arms: Experimental: Supervisor Intervention
Other: Waitlist Control — Control group will receive training following all measurements points to serve as a comparison group
  Arms: Waitlist Control Group

SUMMARY:
The Study for Employment Retention of Veterans (SERVe) is a randomized controlled trial, available exclusively to Oregon employers of veterans. It is designed to develop and scientifically evaluate Veteran-supportive supervisor training (VSST) that may enhance retention of veterans, with the goal of improving workplace culture and general well-being to our service members. The intervention, applied to workplace supervisors, will be measured by experience of veterans, assessing workplace experiences, health, well-being, as well as employees' spouse/partners' family experiences, health and well-being, and workplace outcomes.

DETAILED DESCRIPTION:
The overall goal of the Study for Employment Retention of Veterans (SERVe) study is to improve health and well-being of current and former service members employed in participating Oregon organizations. The SERVe Study seeks to do this by training supervisors to support veteran employees by focusing on a reduction in work-life stress while increasing supportive supervisor behavior.

The SERVe Study proposes that supervisor supportiveness can influence workplace experience, health, and well-being of service members, as well as of their families.

The investigators of the SERVe Study expect positive results for study participants, including reduced stress and increased social support, reduction in negative workplace experiences, and improvement in family well-being outcomes. Longer term, these effects are expected to create a more supportive work environment, which has positive effects on safety, health, well-being, family, and organizational outcomes.

Veteran participants are measured at baseline, three months, and nine months. Veteran spouses are invited to participate as well. Married and cohabitating veterans and their partners are invited to participate in the Daily Family Study (DFS), a 32-day daily diary survey after baseline and at six months.

ELIGIBILITY:
Inclusion Criteria:

* Must have served in the United States Armed Forces since September, 2001
* Must work at least 20 hours per week at a participating organization

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2013-04; Primary Completion 2016-06 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Change in Veteran Supportive Supervisor Behavior as measured by Perry et al.'s (2017) scale | 3 month and 9 months after Baseline assessment
  VSSB as measured by Perry et al.'s (2017) scale, as impacted by the Veteran Supportive Supervisor Training

SECONDARY OUTCOMES:
Change in Work-Family Conflict as assessed by Matthews et al.'s (2010) Work-Family Conflict Scale | 3 and 9 months after baseline assessment
  as assessed by Matthews et al.'s (2010) Work-Family Conflict Scale

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Hammer, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No